CLINICAL TRIAL: NCT04091191
Title: A Single Center, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Tolerability of a Specialized Nutraceutical for Endometriosis
Brief Title: Evaluation of a Nutraceutical for Endometriosis Pain Relief
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Metagenics Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Meta19.01
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specialized nutraceutical (Active Comparator): Specialized nutraceutical formulated in softgel. Participants are instructed to take 2 softgels orally with some water, one before breakfast and one before diner.
  Interventions: Dietary Supplement: Meta19.01
- Placebo (Placebo Comparator): Identical placebo formulated without active ingredients in softgel. Participants are instructed to take 2 softgels orally with some water, one before breakfast and one before diner.
  Interventions: Dietary Supplement: Meta19.01

INTERVENTIONS:
Dietary Supplement: Meta19.01 — A specialized nutraceutical containing plant extracts, vitamins and fish oil

SUMMARY:
Based on the EHP-30 questionnaire, the pain score and general well-being of all patients will be assessed with and without taking a specialized nutraceutical. These patients will be taking continuous oral contraception, for 3 months before inclusion till at least end of the study or not taking any oral contraception at all during the study due to contraindication(s).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed endometriosis and/or Positive NMR
* 18-49y
* Mean pain score >6 on the assessment of pelvic pain (Visual analogue scale)
* Not eligible for surgery in the coming 3 months or had surgery >3 months before inclusion in the study
* >3 months intake of continue oral contraception (Oestrogen/Progesterone) before inclusion or no intake of oral contraception due to contraindication
* Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Planned surgery during study
* <3 month intake of continue oral contraception (Oestrogen/Progesterone) before inclusion
* Chronic inflammatory disease (Chron's disease, Rheumatism,..)
* Pregnancy
* Bariatric surgery
* Malabsorption issues
* Allergy or hypersensitivity to the study product:
* Fish and products thereof: fish oil
* Soybeans and products thereof
* Alcohol or substance abuse
* Start of gonadorelin analogue (ex. Busereline, Gosereline, triptoreline) therapy in the past 6 months
* Intake of other food supplements, including omega 3 and omega 6
* Any other condition which in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Pain relief | 3 months
  pain relief monitored via the Assessment of Pelvic Pain (Visual Analogue scale, VAS) in the Endometriosis Health Profile 30 questions (EHP-30) at baseline and after 3 months of study product intake. The mean of all 3 VAS scales is taken to monitor the evolution of the pain of the subjects. Scores can be given from 0 to 10 with 0 as no pain and 10 as unbearable pain.

SECONDARY OUTCOMES:
Inflammation marker C-reactive protein (CRP) | 3 months
  CRP will be measured at baseline and after 3 months of study product intake. High CRP values (>3mg/L) indicate inflammation while low CRP values (<1 mg/L) indicate no inflammation.
General well-being | 3 months
  The general well-being will be monitored via the Endometriosis Health Profile questionnaire with 30 questions (EHP-30) at baseline and after 3 months of product intake. These scales are transformed into a score from 0 to 100, in which 0 indicates a better health status, while 100 indicates a worse quality of life.
The need for analgesics | 3 months
  The need for analgesics while taking the study product will be monitored via an analgesic diary completed every time the subject takes pain medication. Over 3 months, the total need for analgesics per month will be counted and compared inbetween both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yaacoub Salame, MD, Principal Investigator — CHU Ambroise Paré de Mons
Locations (1):
- CHU Ambroise Paré de Mons, Mons, Hainout, Belgium

IPD SHARING:
Plan to Share IPD: No